CLINICAL TRIAL: NCT05085925
Title: Randomized Intervention Study of Mindfulness-Based Stress-Reduction to Improve the Quality of Life and Immune Regulation in Patients With Crohn's Disease
Brief Title: Mindfulness-Based Stress-Reduction in Patients With Crohn's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Principal Investigator, Dr Doron Schwartz, Senior Physician, Department of Gastroenterology and Hepatology, Soroka University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOR- 0063-20-CTIL; 2018PG-CD005 (Other: The Leona M. and Harry B. Helmsley Charitable Trust)
Record Dates: First submitted 2020-02-18; First posted 2021-10-20 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Crohn's Disease Colon
Keywords: Crohn's Disease; Health-related quality of life; Cognitive behavioral therapy; Mindfulness; Healthcare cost; Immune regulation
MeSH Terms: conditions — Crohn Disease | interventions — Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive behavioral mindfulness intervention at entry (Experimental): Cognitive behavioral mindfulness intervention at entry
  Interventions: Behavioral: Cognitive behavioral mindfulness intervention
- Cognitive behavioral mindfulness intervention after 3 months (Active Comparator): Cognitive behavioral mindfulness intervention after 3 months of wait list
  Interventions: Behavioral: Cognitive behavioral mindfulness intervention after 3-month wait list

INTERVENTIONS:
Behavioral: Cognitive behavioral mindfulness intervention — The group that receives mindfulness-based stress reduction at their entry into the study will have 7 sequential sessions during 3 months, and later have a booster session in month 5
  Arms: Cognitive behavioral mindfulness intervention at entry
Behavioral: Cognitive behavioral mindfulness intervention after 3-month wait list — Wait-list control patients will get no intervention at the start of the study and instead will be contacted by study personal 7 times to care for the patient in order to control for the 7 sessions performed in the intervention group. After three months they will be offered mindfulness-based stress reduction as 8 sequential sessions.
  Arms: Cognitive behavioral mindfulness intervention after 3 months

SUMMARY:
A randomized controlled study which aims to improve the quality of life of Crohn's disease adult patients suffering from mild to moderate level of symptoms. Patients will be randomized to Intervention or Wait-List groups and will undergo eight Cognitive Behavioral and Mindfulness, one on one, sessions with a social worker via SkypeTM. The Intervention group will receive intervention upon recruitment while the Wait-List group will receive the same intervention after 3 months. Clinical, biological and psycho-social data will be collected at four time points over the 12-months of the study.

DETAILED DESCRIPTION:
1. Overall objectives:

   1. Primary outcome: To determine whether mindfulness-based stress reduction will lead to a better health-related quality-of-life by use of three questionnaires:

      • the Crohn's disease specific SIBDQ (Short Inflammatory Bowel Disease Questionnaire, with mean score and 4 subscales: bowel, systemic, social, emotional)
      * SF-12 (MOS Short-Form-12) which is derived from the generic SF-36 used in our previous research (SF-36 measures a Physical Health Summary Score comprised of physical functioning, role-physical, bodily pain and general health, and a Mental Health Summary Score comprised of vitality, role-emotional, social functioning and mental health).
      * EQ-5D (EuroQol questionnaire, for calculation of utility weights)
   2. Secondary outcomes: improvement in mindfulness (FMI, Freiburg Mindfulness Inventory); reduction of stress, anxiety and depression (BSI - Brief Symptom Inventory, GSI - General Severity Index stress measure, MSPSS- Multidimensional Scale of Perceived Social Support, PSS-4 Perceived Stress Scale, LEQ- life events questionnaire); better satisfaction with life (SWLS, Satisfaction with Life Scale); improved family function (FAD, Family Assessment Device); pain reduction (HBI, Harvey-Bradshaw Index of activity of Crohn's disease); less fatigue (FACIT Fatigue Scale); better coping with disease (COPE: Brief Cope Inventory - Brief Coping Operations Preference Enquiry); better performance at work (WPAI, Work Productivity and Activity Impairment) and cost estimation. Significant changes in the scores of these questionnaires, based on our current work comparing P-HBI remission versus active disease, are the following (all are given in points, except WPAI is percent): SIBDQ 6, SWLS 5, FAD 0.15, COPE dysfunctional 2.5, COPE emotion-focused 0.7, COPE problem-focused 0.6, WPAI time missed 14, WPAI percent impairment 29, WPAI work impairment 28, WPAI activity impairment 30, GSI 0.6, BSI anxiety 0.6, BSI depression 0.6. We did not use the SF-12, EQ-5D, MSPSS, PSS-4 and the FACIT Fatigue Scale in our previous research and will look at reports in the literature and our newly acquired data to determine what are significant improvements.
   3. Before and at the end of each intervention session a short assessment of patient's subjective units of distress (SUDS) will be done, as per Wolpe, Joseph (1969), The Practice of Behavior Therapy, New York: Pergamon Press, and the 4 question Short-Form Perceived Stress Scale, as per Warttig et al, J Health Psychology 2013;18:1617-28.
   4. Correlations of psychological measures with demography, economic status, HBI, immune regulation, telomere shortening, fMRI data, changes in composition of microbiota. Change in biophysical parameters as sleep physical activity & pulse rate.
   5. To determine whether the intervention is cost-saving or cost-effective, by prospective monitoring of resource use and indirect costs.
   6. To determine whether the intervention can be given effectively using telemedicine with Skype or alternative software.
   7. To study patient acceptability of the intervention, including recruitment and drop-out rate, and the adherence rate to home practice of the stress reduction measure taught.
2. Expected outcomes

   1. Reduced HBI, improvement of all the psychological measures including both quality-of-life and satisfaction with life, less stress, less fatigue, more use of adaptive coping strategies, with no clear improvements in the control group. Improvement in biophysical parameters as sleep physical activity & pulse rate.
   2. The research will identify the best form of delivering the interventional therapy and if it is cost-saving or cost-effective.
   3. Confirmation of the reliability of measurements of modification of immune regulation mechanisms and telomere length, grey matter thickness and composition of the microbiota.
   4. Glucocorticoid resistance and related laboratory determinations on patients' leukocytes will add to understanding the biological mechanisms associated with stress-induced pathogenic autoimmunity in the patients in a sex-dependent manner. This will add to our understanding the biological mechanisms associated with stress in Crohn's disease.
3. Work plan and methodology

   a. Patient recruitment i. Patients: 200 patients being treated at all the participating hospitals (Soroka Medical Center, Rambam Health Campus, Sheba Medical Center, Rabin Medical Center, Shaare Zedek Medical Center), which all have electronic records of large cohorts of patients with Crohn's disease and by advertising through patient support groups and institutions upon approval. The recruitment of patients will be offered in all the hospitals. Preference will be given to patients who have participated in the previous IIRN study and are now participating in the new IIRN studies proposed by the other hospitals, and those patients in higher risk groups (poorer men, female gender, etc.).

iv. Patients on a fixed dose of corticosteroids and those who received corticosteroid therapy in last 6 months will present a special sub-group on whom the laboratory studies of cortisol and glucocorticoid resistance may differ significantly from patients not on this treatment, but this will have to be verified by measurements in a small sample to determine the magnitude of the effect before a decision to include or exclude these individuals.

v. Patients with change of diagnosis in the course of the study period will be excluded from the final analysis.

vi. Ethical considerations: This protocol will need approval of the Ethics Committee at all hospitals prior to commencement of patient recruitment and access of patient data at these hospitals. A signed informed consent form will be obtained from each participant.

b. Assessment of patient status i. Medical status (HBI) and phenotype. No attempt will be made to modify the patients' treatments.

ii. Psycho-social self-report questionnaires: demography, economic status, SIBDQ, EQ-5D, SF-12, WPAI, SWLS, FACIT, COPE, FAD, BSI, GSI, FMI, MSPSS, PSS-4, LEQ.

iii. Objective outcomes:

1. HBI, CRP, calprotectin, relevant imaging studies (radiology, endoscopy) biophysical parameters as sleep physical activity & pulse rate.
2. Special tests on all or selected sub-sets of patients: immune regulation, telomeres, fMRI, and microbiota.
3. Biophysical parameters as sleep physical activity & pulse rate will be monitored in 30 patients by using commercially available smart watches.

   c. Psycho-social interventions i. The sample size calculation is based on α = 0.05, power = 0.8, SD = 14 (data from our current research) in order to achieve a 6-point change in the SIBDQ (the primary endpoint). Thus, the cohort will consist of 172 patients computer-randomized to two groups; 86 patients with mindfulness-based stress reduction, and 86 wait-list controls that will enter the intervention phase after 3 months. In order to allow for a 15% expected drop-out rate, these recruitment numbers may need to be increased to 200 patients. An equal number of women and men will be recruited at each hospital.

   ii. The group that receives mindfulness-based stress reduction at their entry into the study will have 7 sequential sessions during 3 months, and later have a booster session in month 5. This group will have 4 time points for assessment (see Table, below).

   iii. Wait-list control patients will get no intervention at the start of the study and instead will be contacted by study personal 7 times to care for the patient in order to control for the 7 sessions performed in the intervention group. After three months they will be offered mindfulness-based stress reduction as 8 sequential sessions. The reason for wait-listing is to ensure that there will be a control group to parallel the first 3 months of intervention therapy in the patients getting the therapy from the start. The control group will have the same time points for data assessment as the intervention group.

   iv. All interventions will be individual sessions. v. Patients will be accessed via internet apps such as Skype. vi. Mindfulness-based stress reduction is to be given by specially trained therapists: These are social workers (PhD or Masters candidate level), who have undergone a training session program provided by relevant researchers of this protocol (including clinicians) as well as invited outside psychologists and psychiatrists with specialization in this field.

   vii. Psycho-social, medical and biological data will be collected at the measurement points T1, T2, T3 and T4 (see Table) in all patients. fMRI (to be performed at Soroka Medical Center, without use of contrast) and microbiota studies (stool samples) will be performed on a subset of patients.

   d. Health-care cost i. Direct costs: admissions to hospital, surgery, consultations (primary care physicians, specialists, dieticians, social services) investigations and medications, travel costs to medical facilities.

   ii. Indirect costs: lost workdays, lost productivity, disability payments, travel costs and expenses of escorts.

   e. Immune regulation studies, glucocorticoid resistance in lymphocytes, telomeres i. Blood collections (see Table of events, below) will be performed on consenting patients with Crohn's disease before and after Mindfulness-based stress reduction at 3 time points, as well as in age- and gender-matched consenting healthy volunteer controls (consenting patients without inflammatory diseases attending at the Gastroenterology Department at Soroka Medical Center for screening endoscopies) at one time points.

   ii. Blood will be drawn immunological and telomere studies.

1. Immunology: Blood is sampled twice from 60 Crohn's disease and from 60 controls for isolation of serum and peripheral blood mononuclear cell aliquots at enrollment and after Mindfulness-based stress reduction (provided these patients enter a phase of remission). Serum measures will include plasma C-reactive protein (CRP), ACTH, CBG and sex hormones. Similarly, peripheral blood mononuclear cell will undergo functional immune phenotyping of disease-implicated T cell and B cell subsets and assessments of their glucocorticoid resistance. Glucocorticoid signaling experiments will be performed in purified pro-inflammatory lymphocyte subsets found to exhibit glucocorticoid resistance. Results will be correlated with all other measures in this proposal. Controls for these tests will be matched healthy volunteers. The same tests will be carried out in the controls.

2. Telomere studies in 30 patients with Crohn's disease and 30 controls: by TeloTAGGG™ Telomere Length Assay (Merck). Two blood samples will be needed (see Table of events, below) f. Stool testing - stool samples will be collected at T1 and T2 i. Calprotectin will be measured in the stool at T1 and T2. ii. Microbiota study will be performed on 30 intervention patients and 30 control patients.

g. fMRI - A non-contrast brain MRI will be performed on 30 intervention and 30 control patients at T1 and T2

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate and commit to a one-year process
* Age 18-75 years
* Hebrew-speaking
* Proven diagnosis of mild/moderate Crohn's disease
* At least 3 months post-diagnosis

Exclusion Criteria:

* Crohn's disease that is severe (HBI >16) or in remission (HBI<5)
* Ulcerative colitis, IBD unclassified
* Planned surgery or surgery in last 6 months
* Psychiatric disease
* Psychotropic medication
* Alcohol or drug dependency
* Pregnancy
* Significant or poorly controlled comorbidity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2021-07-16 (Actual)

PRIMARY OUTCOMES:
Change in Crohn's disease specific health-related quality of life | Measured at baseline, 3-months, 6-months, 12-months
  Measured by the Short Inflammatory Bowel Disease Questionnaire (SIBDQ). Range: 10-70; Higher score indicates better quality of life
Change in general health profile | Measured at baseline, 3-months, 6-months, 12-months
  Measured by the Short Form-12 (SF-12); 0-100; Higher scores indicate better quality of life
Change in utility weights | Measured at baseline, 3-months, 6-months, 12-months
  Measured by the EuroQoL (EQ-5D-3L); 0-1; Higher scores indicate higher and better utility weights

SECONDARY OUTCOMES:
Social support | Measured at baseline, 3-months, 6-months, 12-months
  Measured by the Multidimensional Scale of Perceived Social Support: Family, friends and significant other (MSPSS); 1-7; Higher scores indicate better support
Stress, anxiety and depression | Measured at baseline, 3-months, 6-months, 12-months
  Measured by BSI - Brief Symptom Inventory, GSI - General Severity Index stress measure, MSPSS- Multidimensional Scale of Perceived Social Support, PSS-4 Perceived Stress Scale, LEQ- life events questionnaire
Perceived stress | Measured at baseline, 3-months, 6-months, 12-months
  Measured by the Perceived Stress Scale (Pass-4); 0-16; Higher score indicated higher stress
Satisfaction with life | Measured at baseline, 3-months, 6-months, 12-months
  Measured by SWLS, Satisfaction with Life Scale; 5-35; Higher score indicates higher satisfaction with life
Fatigue | Measured at baseline, 3-months, 6-months, 12-months
  Measured by FACIT-Fatigue Scale; 0-52; Higher score indicates better outcome
Pain reduction | Measured at baseline, 3-months, 6-months, 12-months
  Measured by the Harvey-Bradshaw Index (HBI) of activity of Crohn's disease
Coping with disease | Measured at baseline, 3-months, 6-months, 12-months
  Measured by the Brief Coping Operations Preference Enquiry (COPE). HIgher score indicates higher usage of coping strategy
  Problem focus coping strategy (COPE PFS) subscale; 0-24; Higher score means higher use of this efficient mechanism.
  Emotional focused coping strategy (COPE EFS) subscale; 10-40; Higher score means higher use of this controversial mechanism.
  Dysfunctional focus coping strategy (COPE DFS) subscale; 12-48; Higher score means higher use none-efficient mechanism.
Performance at work | Measured at baseline, 3-months, 6-months, 12-months
  Measured with WPAI, Work Productivity and Activity Impairment
Resource utilization and healthcare costs | Measured at baseline, 3-months, 6-months, 12-months
  Patient self report
Mindfulness | Measured at baseline, 3-months, 6-months, 12-months
  Self report of patient's mindfulenss level, measured with FMI (Freiburg Mindfulness Inventory); 14-56; higher score indicates a greater self percived mindfulness level
Family Support | Measured at baseline, 3-months, 6-months, 12-months
  Self report of patient's family support, measured with FAD (Family Assessment Device);

CONTACTS AND LOCATIONS:
Overall Officials: Ganit Goren, MA, Study Director — Ben-Gurion University of the Negev
Locations (1):
- Soroka University Medical Center, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391
- [Derived] Goren G, Schwartz D, Friger M, Sergienko R, Monsonego A, Slonim-Nevo V, Greenberg D, Odes S, Sarid O. Gender Differences in Coping Strategies and Life Satisfaction Following Cognitive-Behavioral and Mindfulness-Based Intervention for Crohn's Disease: A Randomized Controlled Trial. J Clin Med. 2025 Feb 26;14(5):1569. doi: 10.3390/jcm14051569. PMID 40095500